CLINICAL TRIAL: NCT02825264
Title: STAR-LIFE Registry: STARflo Glaucoma Implant Clinical Experience Program in a Real-World Patient Population
Brief Title: STAR-LIFE Registry: STARflo Glaucoma Implant Clinical Experience Program
Status: Active, not recruiting | Type: Observational
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISM03
Record Dates: First submitted 2016-06-20; First posted 2016-07-07 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Open Angle Glaucoma
Keywords: Glaucoma Drainage Device; STARflo
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STARflo: Patients who have been implanted with STARflo implant
  Interventions: Device: STARflo Implant

INTERVENTIONS:
Device: STARflo Implant — All patients who have been implanted with STARflo implant from 2011 will be offered to participate to this data collection

SUMMARY:
STARflo is a novel suprachoroidal Glaucoma Drainage Device (GDD), bleb-free, exhibiting anti-fibrotic properties. Release of this CE Marked implant has been limited to leading Glaucoma Centers in Europe.

DETAILED DESCRIPTION:
This Clinical Experience Program is being initiated to expand the surgical and clinical practice knowledge about the use of STARflo for reducing intraocular pression (IOP) in patients suffering from open angle glaucoma in a real world population of patients.

This program is designed to be an international multicenter observational study.

Patient data may be collected retrospectively and/or prospectively for up to 5 years after surgery.

The aim of this program is to document the patient's benefit following implantation of the STARflo implant in a real-word patient population, to learn about surgical practices and to collect data to support future cost-effectiveness analysis.

ELIGIBILITY:
Inclusion criteria:

* Patients suffering from open angle glaucoma or some case of narrow angle glaucoma who have been implanted with STARflo implant from 2011
* Patients who have signed a Data Release form

Exclusion criteria:

* Patients who did not sign a Data Release form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from open angle glaucoma or some case of narrow angle glaucoma who have been implanted with STARflo.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of intraocular pressure (IOP) | at 12 Months
  IOP reduction compared after 12 months compared to baseline IOP

SECONDARY OUTCOMES:
Occurence of Ocular Adverse Events | up to 60 Months after surgery
  to record and document all complications and Adverse Events/Adverse Device Effects occurred during and after surgery
Reduction of intraocular pressure (IOP) over time | at 6, 24, 36, 48 and 60 Months
  IOP reduction compared after 6, 24, 36, 48 and 60 months compared to baseline IOP
Reduction of IOP lowering medication | at 6, 12, 24, 36, 48 and 60 Months
  Reduction of IOP lowering medication intake compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — Sponsor Representative
Locations (9):
- Bât. BC-3 OPHTALMOLOGIE - POLICLINIQUE C.H.U., Liège, Belgium
- France (2):
  - Hospital de la Croix-Rousse, Lyon
  - CHNO des Quinze-Vingts, Paris
- Germany (4):
  - St. Johannes Hospital Dortmund, Dortmund
  - Universitäts-Augenklinik Heidelberg, Heidelberg
  - Klinikum der Universität München, München
  - Augenklinik Universitätsmedizin Rostock, Rostock
- Elisabeth Academic Hospital, Sopron, Hungary
- Hospital Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided